CLINICAL TRIAL: NCT02340949
Title: Induction FOLFOX With or Without Aflibercept Followed by Chemoradiation in High Risk Locally Advanced Rectal Cancer. Phase II Randomized, Multicenter, Open Label Trial
Brief Title: Induction FOLFOX With or Without Aflibercept Followed by Chemoradiation in High Risk Locally Advanced Rectal Cancer
Acronym: RIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol Multidisciplinario del Cancer Digestivo (Other)
Collaborators: Pivotal S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEMCAD-1402
Record Dates: First submitted 2015-01-09; First posted 2015-01-19 (Estimated); Results first posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — aflibercept; Fluorouracil; Oxaliplatin; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mFOLFOX6 + Aflibercept (Experimental): - mFOLFOX-6 scheme: 5-Fluoruracil [5-FU], oxaliplatin and leucovorin will be administered intravenously once every 14 days according to mFOLFOX-6 scheme:
  Day 1: Oxaliplatin 85 mg/m² IV infusion in 250-500 mL and leucovorin 200 mg/m² IV, both over two hours, followed by 5-FU 400 mg/m² IV bolus and a 46 h infusion of 5-FU 2400 mg/m².
  - Aflibercept, will be administered intravenously (I.V.) at doses of 4 mg/Kg on Day 1 every 14 days. Aflibercept will be supplied to sites by the study Sponsor as 4 ml vials at a concentration of 25 mg/ml.
  Treatment will continue until six cycles are administered unless unacceptable toxicity or progression occurs.
  Interventions: Drug: Aflibercept; Drug: 5-Fluoruracil; Drug: Oxaliplatin; Drug: Leucovorin
- mFOLFOX6 (Active Comparator): - mFOLFOX-6 scheme: 5-Fluoruracil [5-FU], oxaliplatin and leucovorin will be administered intravenously once every 14 days according to mFOLFOX-6 scheme:
  Day 1: Oxaliplatin 85 mg/m² IV infusion in 250-500 mL and leucovorin 200 mg/m² IV, both over two hours, followed by 5-FU 400 mg/m² IV bolus and a 46 h infusion of 5-FU 2400 mg/m².
  Treatment will continue until six cycles are administered unless unacceptable toxicity or progression occurs.
  Interventions: Drug: 5-Fluoruracil; Drug: Oxaliplatin; Drug: Leucovorin

INTERVENTIONS:
Drug: Aflibercept — Administered I.V. at doses of 4 mg/Kg on Day 1 every 14 days. It will be supplied to sites by Sponsor as 4 ml vials at a concentration of 25 mg/ml
  Other Names: ZALTRAP
  Arms: mFOLFOX6 + Aflibercept
Drug: 5-Fluoruracil — Once every 14 days. Day 1: 400 mg/m2 I.V. bolus and a 46 h infusion of 5-FU 2400 mg/m2
  Other Names: 5-FU
Drug: Oxaliplatin — Once every 14 days. Day 1: 85 mg/m2 I.V. infusion in 250-500 mL, over two hours, followed by 5-FU
  Other Names: Any marketed
Drug: Leucovorin — Once every 14 days. Day 1: 200 mg/m2 I.V., over two hours, followed by 5-FU
  Other Names: Any marketed

SUMMARY:
This trial compares induction treatment with FOLFOX with or without aflibercept in a high risk population selected by MRI, prior to receiving standard chemoradiation (capecitabine combined with 50.4 Gy in 28 days) and surgery, in order to evaluate the efficacy in terms of pathologic complete response (pCR).

DETAILED DESCRIPTION:
This is a randomized trial comparing induction treatment with FOLFOX with or without aflibercept in a high risk population selected by MRI, prior to receiving standard chemoradiation (capecitabine combined with 50.4 Gy in 28 days) and surgery. Once it is confirmed that the subjects fulfill the eligibility criteria (MRI-defined high risk RC), and have signed the informed consent, a central review will be requested to confirm clinical stage, and then they will be randomized to receive mFOLFOX6 + Aflibercept or mFOLFOX6 (without Aflibercept).

Random assignment of treatment will be stratified by T3 versus T4 stage. All the patients enrolled in the study will receive one cycle of study medication (mFOLFOX6 with or without aflibercept) every 14 days for six cycles, unless unacceptable toxicity or progression is detected. After this treatment, patients will receive standard chemo-radiotherapy (CT/RT) (capecitabine 825 mg/m2 twice daily combined with a total dose of 50.4 Gy in 28 days) followed by surgery, provided they have not progressed.

Patients with progression disease during the treatment phase will be withdrawn from the study and will receive their treatment according to the investigator's judgment. If a patient withdraws consent and refuses to receive further treatment, the patient must be followed up for 3 years from randomization or until progression, to evaluate disease-free survival. If a patient withdraws consent and refuses to continue in the study, the follow-up evaluations must be discontinued.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent, and willing and able to comply with protocol requirement;
2. Male or female subjects with rectal cancer ≥18 and <70 years of age;
3. High risk MRI-defined operable rectal cancer (with an inferior margin no more than 12 cm above the anal verge as assessed by MRI). Presence of at least 1 of the following on high resolution, thin-slice MRI (3 mm):

   Middle Third Tumors
   * mr T3

     1. Extramural vascular invasion (EMVI) positive
     2. Extramural extension > 5 mms into perirectal fat
     3. Mesorectal fascia (MRF) threatened or involved*
   * mr T4***

   Distal Third Tumors (≤5 cm from anal verge)
   * mr T3 tumor at or below levators
   * T4 as above N2**

     * tumor or lymph node < 1 mm from the mesorectal fascia **≥4 lymph nodes in the mesorectum showing morphological signs on MRI indicating metastatic disease. ≥4 nodes, whether enlarged or not, with a rounded, homogeneous appearance is thus not sufficient.

       * T4a: overgrowth to an adjacent organ or structure or T4b: peritoneal involvement.
4. Histologically confirmed adenocarcinoma of the rectum. All other histological types are excluded;
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤1;
6. Hematological status: neutrophils (ANC) ≥1.5x109/L; platelets ≥100x109/L; hemoglobin ≥9g/dL;
7. Adequate renal function: serum creatinine level <1.5 x upper limit of normality (ULN);
8. Adequate liver function: serum bilirubin ≤1.5 x ULN, alkaline phosphatase <5x ULN, AST/ALT < 3 x ULN;
9. Proteinuria <2+ (dipstick urinalysis) or ≤1g/24hour;
10. Regular follow-up feasible;
11. For female patients of childbearing potential, negative serum pregnancy test within 1 week (7 days) prior to starting study treatment;
12. Female patients must commit to using reliable and appropriate methods of contraception until at least three months after the end of study treatment (when applicable). Male patients with a partner of childbearing potential must agree to use contraception in addition to having their partner use another contraceptive method during the trial.

Exclusion Criteria:

1. Prior treatment with aflibercept;
2. History or evidence upon physical examination of metastasis;
3. Uncontrolled hypercalcemia;
4. Pre-existing permanent neuropathy (NCI grade ≥2);
5. Uncontrolled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg), or history of hypertensive crisis, or hypertensive encephalopathy;
6. Concomitant protocol unplanned antitumor therapy (e.g. chemotherapy, molecular targeted therapy, immunotherapy);
7. Treatment with any other investigational medicinal product within 28 days prior to study entry;
8. Other concomitant or previous malignancy, except: i/ adequately treated in-situ carcinoma of the uterine cervix, ii/ basal or squamous cell carcinoma of the skin, iii/ cancer in complete remission for >5 years;
9. Any other serious and uncontrolled non-malignant disease, major surgery or traumatic injury within the last 28 days;
10. Pregnant or breastfeeding women;
11. Patients with known allergy to any excipient to study drugs;
12. History of myocardial infarction and/or stroke within 6 months prior to randomization; Previous history of stable angina, uncontrolled arrhythmia, and acute coronary syndrome even if controlled with medication or with myocardial infarction within the last 12 months.
13. Bowel obstruction.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-01; Primary Completion 2019-07-15 (Actual); Study Completion 2020-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Fernández-Martos, MD, Study Director — Fundación Instituto Valenciano de Oncología; Antonieta Salud Salvia, MD, Principal Investigator — Hospital Universitari Arnau de Vilanova de Lleida; Carles Pericay Pijaume, MD, Principal Investigator — Hospital de Sabadell - Parc Taulí; Clara Montagut, MD, Principal Investigator — Hospital del Mar; Joan Maurel Santasusana, MD, Principal Investigator — Hospital Clinic i provincial de Barcelona; Vicente Alonso Orduña, MD, Principal Investigator — Hospital Miguel Servet; Ruth Vera García, MD, Principal Investigator — Complejo Hospitalario de Navarra; Javier Gallego Plazas, MD, Principal Investigator — Hospital General Universitario de Elche; Núria Rodríguez Salas, MD, Principal Investigator — Hospital Universitario La Paz; Antonio Cubillo, MD, Principal Investigator — Hospital Universitario Madrid Sanchinarro (CIOCC); Bertomeu Massuti, MD, Principal Investigator — Hospital General Universitario de Alicante; Ferrán Losa, MD, Principal Investigator — Hospital de Sant Joan Despí Moisés Broggi; Miguel Nogué, MD, Principal Investigator — Hospital General de Granollers; Jaume Capdevila, MD, Principal Investigator — Hospital Universitari Vall d'Hebrón; Isabel Busquier, MD, Principal Investigator — Consorcio Hospitalario Provincial de Castellón; Inma Guash Jordan, MD, Principal Investigator — Fundación Althaia Manresa; Laura Layos Romero, MD, Principal Investigator — Hospital Universitari Germans Trias i Pujol de Badalona; Marta Martín-Richard, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Rocio García Carbonero, MD, Principal Investigator — Hospital Universitario 12 de Octubre; Carlos López López, MD, Principal Investigator — Hospital Universitario Marqués de Valdecilla

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandez-Martos C, Pericay C, Losa F, Garcia-Carbonero R, Layos L, Rodriguez-Salas N, Martin-Richard M, Alonso-Orduna V, Vera R, Gallego J, Capdevila J, Salud A, Nogue M, Maurel J, Guash I, Montagut C, Lopez C, Macias I, Jain RK, Garcia-Albeniz X. Effect of Aflibercept Plus Modified FOLFOX6 Induction Chemotherapy Before Standard Chemoradiotherapy and Surgery in Patients With High-Risk Rectal Adenocarcinoma: The GEMCAD 1402 Randomized Clinical Trial. JAMA Oncol. 2019 Nov 1;5(11):1566-1573. doi: 10.1001/jamaoncol.2019.2294. PMID 31465088

RESULTS

PARTICIPANT FLOW:
Groups:
- mFOLFOX6 + Aflibercept: - mFOLFOX-6 scheme: 5-Fluoruracil [5-FU], oxaliplatin and leucovorin will be administered intravenously once every 14 days according to mFOLFOX-6 scheme:
  Day 1: Oxaliplatin 85 mg/m² IV infusion in 250-500 mL and leucovorin 200 mg/m² IV, both over two hours, followed by 5-FU 400 mg/m² IV bolus and a 46 h infusion of 5-FU 2400 mg/m².
  - Aflibercept, will be administered intravenously (I.V.) at doses of 4 mg/Kg on Day 1 every 14 days. Aflibercept will be supplied to sites by the study Sponsor as 4 ml vials at a concentration of 25 mg/ml.
  Treatment will continue until six cycles are administered unless unacceptable toxicity or progression occurs.
  Aflibercept: Administered I.V. at doses of 4 mg/Kg on Day 1 every 14 days. It will be supplied to sites by Sponsor as 4 ml vials at a concentration of 25 mg/ml
  5-Fluoruracil: Once every 14 days. Day 1: 400 mg/m2 I.V. bolus and a 46 h infusion of 5-FU 2400 mg/m2
  Oxaliplatin: Once every 14 days. Day 1: 85 mg/m2 I.V. infusion in 250-500 mL, over two hours, followed by 5-FU
  Leucovorin: Once every 14 days. Day 1: 200 mg/m2 I.V., over two hours, followed by 5-FU
- mFOLFOX6: - mFOLFOX-6 scheme: 5-Fluoruracil [5-FU], oxaliplatin and leucovorin will be administered intravenously once every 14 days according to mFOLFOX-6 scheme:
  Day 1: Oxaliplatin 85 mg/m² IV infusion in 250-500 mL and leucovorin 200 mg/m² IV, both over two hours, followed by 5-FU 400 mg/m² IV bolus and a 46 h infusion of 5-FU 2400 mg/m².
  Treatment will continue until six cycles are administered unless unacceptable toxicity or progression occurs.
  5-Fluoruracil: Once every 14 days. Day 1: 400 mg/m2 I.V. bolus and a 46 h infusion of 5-FU 2400 mg/m2
  Oxaliplatin: Once every 14 days. Day 1: 85 mg/m2 I.V. infusion in 250-500 mL, over two hours, followed by 5-FU
  Leucovorin: Once every 14 days. Day 1: 200 mg/m2 I.V., over two hours, followed by 5-FU
Period: Overall Study
Arm/Group | mFOLFOX6 + Aflibercept | mFOLFOX6
Started | 115 | 65
Completed (Completed the treatment as per protocol) | 99 | 61
Not Completed | 16 | 4
Not completed — Adverse Event | 4 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Progression disease | 6 | 2
Not completed — Death | 3 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | mFOLFOX6 + Aflibercept | mFOLFOX6 | Total
Number analyzed (Participants) | 115 | 65 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years, expressed as "Mean (Standard Deviation)"
  years | 58.4 (10.4) | 62.2 (9.2) | 59.7 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 26 | 64
  Male | 77 | 39 | 116
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Country of recruitment
  Participants
    Spain | 115 | 65 | 180
Clinical stage Tumor-nodes-metastasis (TNM) [Count of Participants; unit: Participants] — TNM clinical stage assessed by magnetic resonance (mr). The T refers to the size and extent of the main tumor.
  Categories assessed by mr:
  T2: limited to bowel wall T3: beyond muscularis propia T3A: <1 mm beyond muscularis propia T3B: 1-5 mm beyond muscularis propia T3C: 5-15 mm beyond muscularis propia T4: involvement peritoneal reflection T4A: involvement peritoneal reflection T4B: ingrowth in organ
  Participants
    Mising | 1 | 1 | 2
    mrT2 | 1 | 0 | 1
    mrT3 | 17 | 12 | 29
    mrT3B | 8 | 8 | 16
    mrT3A | 1 | 0 | 1
    mrT3C | 47 | 22 | 69
    mrT3D | 7 | 4 | 11
    mrT4 | 9 | 6 | 15
    mrT4A | 16 | 7 | 23
    mrT4B | 8 | 5 | 13
Count of Patients Which Had a Baseline Clinical Stage TNM Nodes (n2) [Count of Participants; unit: Participants] — Used to describe regional lymph node involvement of the tumor. N0 indicates no regional nodal spread, while N1-N3 indicates some degree of nodal spread, with a progressively distal spread from N1 to N3.
  Participants | 115 | 65 | 180
Location [Count of Participants; unit: Participants] — Location of primary tumor in the rectum.
  Participants
    Distal | 30 | 18 | 48
    Middle | 84 | 46 | 130
    Missing | 1 | 1 | 2
Histology [Count of Participants; unit: Participants] — Type of tumor cell composition found by histopathology analysis.
  Participants
    Adenocarcinoma | 115 | 65 | 180
    other | 0 | 0 | 0
Mesorectal Fascia (FMR) [Count of Participants; unit: Participants] — Distance from tumor to mesorectal fascia grouped in two categories depending on the distances: close (distance <=1 mm) or distal (NR).
  Participants
    FMR + (distance <=1 mm) | 68 | 37 | 105
    NR | 47 | 28 | 75
EMVI score [Count of Participants; unit: Participants] — Extramural vascular invasion (EMVI) is the direct invasion of a blood vessel (usually a vein) by a tumor. In rectal cancer, this can occur on a macroscopic level and be detected on staging MRI. It is a significant prognostic factor, being a predictor of haematogenous spread. Score range from 0 to 4. Higher score means higher risk of distant metastasis.
  Participants
    Score 0/1/2 | 60 | 34 | 94
    Score 3/4 | 55 | 31 | 86

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving Pathologic Complete Response (pCR).
Description: The number of patients achieving pCR after induction therapy with mFOLFOX6 +/- aflibercept followed by chemotherapy (CT)/radiotherapy (RT). pCR will be defined as the absence of viable tumor cells in the primary tumor and in the lymph nodes (T0N0)
Time Frame: From baseline until 2 years and 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | mFOLFOX6 + Aflibercept | mFOLFOX6
Number analyzed (Participants) | 115 | 65
Participants
  Yes | 25 | 9
  No | 90 | 56

2. Secondary Outcome: Number of Patients Achieving Pathological Parameters of Efficacy: R0 Resection, Tumor Regression Grade, and Circular Radial Margin Rate
Description: R0 resection is defined as complete tumor removal, and correlates with good prognosis.
  Tumor regression grade (TRG) is defined as presence of residual tumor after preoperative therapy. This was assessed by magnetic resonance imaging (MRI) according to the 5-point regression grading scale established by Mandard: TRG1 (complete response with no residual cancer), TRG2 (rare residual cancer), TRG3 (fibrosis outgrowing residual cancer), TRG4 (residual cancer outgrowing fibrosis) and TRG5 (absence of regression).
  Circular Radial Margin (CRM) is defined as the distance from the margin of normal tissue to the edge of tumor tissue in the resected primary tumor the measured by histopathology study after surgery. A margin of ≤1 mm is considered to be a negative prognostic factor for local recurrence.
Time Frame: From baseline until 2 years and 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | mFOLFOX6 + Aflibercept | mFOLFOX6
Number analyzed (Participants) | 115 | 65
Participants
  R0 rate: Yes | 101 | 60
  R0 rate: No | 2 | 2
  R0 rate: Not available | 12 | 3
  TRG1-2: Yes | 59 | 30
  TRG1-2: No | 56 | 35
  TRG1-2: Not available | 0 | 0
  CRM ≤ 1: Yes | 3 | 3
  CRM ≤ 1: No | 96 | 56
  CRM ≤ 1: Not available | 16 | 6

3. Secondary Outcome: Number of Participants With Significant MRI Changes Post Intervention, as Defined by T Downstaging
Description: Tumor size is assessed by MRI to determine the T stage. T Downstaging: defined as a lower pathologic T stage compared to pre-treatment T stage.
Time Frame: From baseline until 2 years and 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | mFOLFOX6 + Aflibercept | mFOLFOX6
Number analyzed (Participants) | 115 | 65
Participants
  Yes | 68 | 46
  No | 47 | 19

4. Secondary Outcome: Number of Patients Reporting Adverse Events (AEs)
Description: The safety and tolerability of the study therapy were assessed by means of AEs and changes in laboratory data. AEs were coded and evaluated using the NCI-CTCAE v4.0 toxicity criteria (if NCI-CTCAE are not applicable, MedDRA was used).
Time Frame: From baseline until 2 years and 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | mFOLFOX6 + Aflibercept | mFOLFOX6
Number analyzed (Participants) | 115 | 65
Participants
  At least one AE: Yes | 115 | 65
  At least one AE: No | 0 | 0
  At least one Grade 3-4 AE: Yes | 83 | 31
  At least one Grade 3-4 AE: No | 32 | 34
  At least one AE that lead to treatment discontinuation: Yes | 20 | 4
  At least one AE that lead to treatment discontinuation: No | 95 | 61
  At least one AE that lead to death: Yes | 3 | 0
  At least one AE that lead to death: No | 112 | 65
  At least one Serious Adverse Event (SAE): Yes | 45 | 16
  At least one Serious Adverse Event (SAE): No | 70 | 49
  At least one treatment-related AE: Yes | 105 | 59
  At least one treatment-related AE: No | 10 | 6
  At least one treatment-related AE Grade 3-4: Yes | 64 | 17
  At least one treatment-related AE Grade 3-4: No | 51 | 48
  At least one treatment-related AE that led to death: Yes | 0 | 0
  At least one treatment-related AE that led to death: No | 115 | 65
  At least one treatment-related AE that led to permanent treatment discontinuation: Yes | 17 | 3
  At least one treatment-related AE that led to permanent treatment discontinuation: No | 98 | 62
  At least one treatment-related Serious Adverse Event (SAE): Yes | 25 | 3
  At least one treatment-related Serious Adverse Event (SAE): No | 90 | 62

5. Secondary Outcome: Number of Patients Reporting Surgical Complications
Description: Surgical complications will be assessed by means of AEs reported during 30 days post surgery.
Time Frame: From surgical intervention up to 30 days post-surgery, within a general time frame of 2 years and 2 months per study protocol
Measure: Count of Participants; unit: Participants
Arm/Group | mFOLFOX6 + Aflibercept | mFOLFOX6
Number analyzed (Participants) | 115 | 65
Participants
  Postoperative AEs: Yes | 3 | 1
  Postoperative AEs: No | 112 | 64
  Postoperative AEs Grade 3-4: Yes | 2 | 0
  Postoperative AEs Grade 3-4: No | 113 | 65
  Complications: Yes | 60 | 30
  Complications: No | 55 | 35
  Anastomosis fistula: Yes | 4 | 1
  Anastomosis fistula: No | 111 | 64
  wound infection: Yes | 5 | 5
  wound infection: No | 110 | 60
  intraabdominal infection: Yes | 10 | 1
  intraabdominal infection: No | 105 | 64
  Stoma complications: Yes | 2 | 0
  Stoma complications: No | 113 | 65
  Reoperation: Yes | 9 | 5
  Reoperation: No | 106 | 60

6. Secondary Outcome: Disease Free Survival (DFS) Rate at 3 Years
Description: DFS rate is defined as the percentage of participants without local recurrences at 3-years post study treatment. Here we report the DFS rate at 3-years after completing the Study treatment.
Time Frame: At 3 years after study treatment completion, within a general time frame of 5 years and two months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | mFOLFOX6 + Aflibercept | mFOLFOX6
Number analyzed (Participants) | 115 | 65
percentage of participants | 75.2 [66.1 to 82.2] | 81.5 [69.8 to 89.1]

ADVERSE EVENTS:
Time Frame: From Baseline to study completion, within an general time frame of 3 years per study protocol
Description: For the statistical tables, adverse events have been coded according to the Medical Dictionary of Regulatory Activities (MedDRA 20.1) system. Their intensity has been coded by (NCI-CTCAE) v4.0 toxicity criteria.
  The safety and tolerability of the study therapy were assessed by means of AEs and changes in laboratory data that were reported in the AEs page.
  Grade 3 or higher AEs were reported as serious. All the grade 1 and 2 as non serious.
Arm/Group | mFOLFOX6 + Aflibercept | mFOLFOX6
All-Cause Mortality (participants affected / at risk) | 12/115 | 7/65
Serious Adverse Events (participants affected / at risk) | 45/115 | 16/65
Other Adverse Events (participants affected / at risk) | 115/115 | 65/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mFOLFOX6 + Aflibercept (N=115) | mFOLFOX6 (N=65)
Asthenia (General disorders) | 2 | 0
Peripheral neuropathy (Nervous system disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 8 | 4
Mucosal inflamation (Gastrointestinal disorders) | 4 | 0
Nausea (General disorders) | 0 | 1
Hypertension (Vascular disorders) | 34 | 2
Neutropenia (Blood and lymphatic system disorders) | 25 | 14
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 0
Abdominal pain (General disorders) | 1 | 0
Dysphonia (General disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Proctalgia (Gastrointestinal disorders) | 1 | 1
Rectal hemorrage (Gastrointestinal disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 0
Stomatitis (Infections and infestations) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mFOLFOX6 + Aflibercept (N=115) | mFOLFOX6 (N=65)
Asthenia (General disorders) | 65 | 38
Peripheral neuropathy (Nervous system disorders) | 48 | 30
Diarrhoea (Gastrointestinal disorders) | 42 | 22
Mucosal inflamation (Gastrointestinal disorders) | 48 | 14
Nausea (General disorders) | 37 | 23
Hypertension (Vascular disorders) | 22 | 3
Neutropenia (Blood and lymphatic system disorders) | 14 | 4
Vomiting (Gastrointestinal disorders) | 21 | 13
Decrease apetite (Gastrointestinal disorders) | 25 | 9
Dysaesthesia (Nervous system disorders) | 15 | 10
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 13 | 8
Abdominal pain (General disorders) | 16 | 5
Constipation (Gastrointestinal disorders) | 13 | 9
Paraesthesia (Nervous system disorders) | 11 | 11
Dysphonia (General disorders) | 19 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 7
Proctalgia (Gastrointestinal disorders) | 11 | 6
Rectal hemorrage (Gastrointestinal disorders) | 14 | 3
Pyrexia (General disorders) | 14 | 4
Dysgeusia (General disorders) | 11 | 8
stomatitis (Infections and infestations) | 14 | 3
Musculoesqueletal pain (General disorders) | 11 | 7
Epistaxis (Vascular disorders) | 17 | 1
cystitis (Infections and infestations) | 9 | 7
Anemia (Blood and lymphatic system disorders) | 6 | 7
Aphonia (General disorders) | 14 | 0
Upper abdominal pain (General disorders) | 10 | 3
Fatigue (General disorders) | 7 | 5
Anal inflammation (Gastrointestinal disorders) | 10 | 0
Rectal tenesmus (Gastrointestinal disorders) | 8 | 1
Headache (General disorders) | 8 | 1

LIMITATIONS AND CAVEATS:
There are no overall limitations and caveats. In detail: There were 6 patients that received treatment doses that did not matched protocol specifications. These were notified as protocol major deviations to the competent authorities and ethics committees. The effect of these deviations on results is not significant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-09): https://cdn.clinicaltrials.gov/large-docs/49/NCT02340949/Prot_SAP_000.pdf